CLINICAL TRIAL: NCT05551494
Title: Urinary Concentration of Phthalate Metabolites in Women With and Without Endometriosis: a Case-control Study
Brief Title: Urinary Concentration of Phthalate Metabolites in Women With and Without Endometriosis
Acronym: FTALATENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Direzione Ginecologia, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 2706
Record Dates: First submitted 2022-08-23; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis
Keywords: phthalates; urinary biomarkers; endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis group: Cases will include women aged 18-45 with a surgical diagnosis of endometriosis in the previous 24 months or with a current nonsurgical diagnosis of endometriosis who report having lived in the past ten years in the Lombardy area. At study entry, we will collect urinary sample.
  Interventions: Diagnostic Test: Urinary sample
- Control group: Control group are women aged 18-45 attending our outpatient clinic for periodical gynaecological care, contraception, or cervical cancer screening programme, and without a previous clinical or surgical diagnosis of endometriosis who report having lived in the past ten years in the Lombardy area. At study entry, we will collect urinary sample.
  Interventions: Diagnostic Test: Urinary sample

INTERVENTIONS:
Diagnostic Test: Urinary sample — At study entry, we will collect urinary samples from women. Participants will be asked with an interview on demographic and lifestyle characteristics, health-related behaviours, the existence and duration of infertility, medical history, and history of hormonal or surgical treatments for endometriosis. Pain symptoms will be evaluated through a 10 cm long one-dimensional visual-analogue scale (VAS).
  In addition, women will be asked to report about their habits about consumption of plastic

SUMMARY:
Exposure to endocrine-disrupting chemicals can considerably affect female reproductive system. Exposure can occur in living environments and in specific workplaces in which these substances are produced or used. Among endocrinedisrupting chemicals, phthalates, dialkyl esters or alkyl aryl esters of orthophthalic acid (1,2-dicarboxylic acid) represent a group of structurally similar molecules, widely used in industry since 1930 in numerous manufacture processes, mainly as a plasticizer.

These substances present dangerous characteristics, particularly associated with reproductive toxicity, and their xenoestrogenicity led some authors to evaluate a possible involvement in the aetiology of endometriosis.

In this proposed study the investigators aim to clarify a potential association between endometriosis and phthalates exposure.

Women with a diagnosis of endometriosis will be recruited as "cases" while women without endometriosis as "controls". An "ad hoc" questionnaire will be administered to the patient to collect the necessary information on the characteristics of endometriosis as well as their lifestyle and work habits.

The biological monitoring will be carried out measuring the urinary levels of phthalate metabolites. In order to produce reliable data and to reduce the possible contamination caused by the contact with plastic materials, samples will be analyzed by High Performance Liquid Chromatography/Tandem Mass Spectrometry (HPLC-MS/MS).

A statistical elaboration of the data will clarify possible identifiable risk factors and associations with specific clinical situations.

The investigators expect that women with endometriosis may present higher levels of phthalates compared with women without the disease. In particular, the investigators hypothesize that women with the most severe form of the disease [i.e. deep infiltrating endometriosis (DIE)] may present the highest levels. These study findings will provide valuable suggestions for developing effective strategies to prevent endometriosis.

DETAILED DESCRIPTION:
Exposure to phthalates can considerably affect female reproductive system. Recent evidence suggests that one of the diseases related to the high concentration of phthalate metabolites in biological fluids might be endometriosis.

This case-control study aims to evaluate the relationship between endometriosis and phthalates exposure through biomarkers analysis in urine. The investigators hypothesize that women with endometriosis, particularly those with deep infiltrating forms (i.e. the most severe form of the disease), will show higher urinary phthalate metabolites compared to women with ovarian/peritoneal forms and those without endometriosis. When deep lesions and ovarian lesions co-existed, the woman will be included in the deep infiltrating subgroup, as the former lesions are considered more severe than the latter ones.

The identification of a possible environmental risk, such as the exposure to phthalates, could allow the implementation of preventive measures aimed at reducing the exposure to such contaminants. Moreover, clinical data obtained may contribute to a better understanding of the etiology and the pathophysiology of endometriosis.

The main objective of the present study is to evaluate the levels of exposure to phthalates of a female population with endometriosis and to understand if it differs significantly from a population of women without the disease.

Identifying a possible relationship between urinary phthalates metabolite concentrations and the risk of endometriosis could represent a valuable tool for implementing specific preventive measures, especially in the workplace.

The results of our case-control study aim to shed more light on the potential association between endometriosis and phthalate exposure, specifically in the Italian context.

Secondary objectives include:

1. to evaluate potential variations in urinary phthalate metabolite levels in women with different phenotypes of the disease: peritoneal endometriosis, ovarian endometriosis, deep infiltrating endometriosis.
2. to evaluate potential variations in the levels of urinary phthalate metabolite in endometriosis patients in relation to the presence and levels of pain symptoms (dysmenorrhea, chronic pelvic pain, deep dyspareunia) and/or infertility.

The causality study will try to identify possible routes of exposure in everyday life and/or working environments, which could represent a possible source of risk. The results could identify work context in which health risks for women could be highly diversified from those for men. This identification could support the competent doctors in defining health surveillance protocols for specific sectors.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis group are women aged 18-45 with a diagnosis of endometriosis who report having lived in the past ten years in the Lombardy area.
* Control group are women aged 18-45 who do not have endometriosis who report having lived in the past ten years in the Lombardy area.

Exclusion Criteria:

* Pregnancy
* Uterine fibroids, gynecological cancers
* Renal, hepatic, cardiovascolar disease, diabetes or high blood pressure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study will be recruited women with or without endometriosis, aged 18-45 years who have lived in the last 10 years in the Lombardy area. Will be excluded women with uterine fibroids, gynecological cancers or renal, hepatic, cardiovascular disease, diabetes or high blood pressure
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate urinary concentration of phthalates | 24 months
  The main objective of the present study is to evaluate the levels of exposure to phthalates of a female population with endometriosis and to understand if it differs significantly from a population of women without the disease. Identifying a possible relationship between urinary phthalates metabolite concentrations and the risk of endometriosis could represent a valuable tool for implementing specific preventive measures, especially in the workplace

SECONDARY OUTCOMES:
Variations in urinary concentration phthalate metabolite levels in women with different phenotypes of the disease | 24 months
  To evaluate potential variations in urinary phthalate metabolite levels in women with different phenotypes of the disease: peritoneal endometriosis, ovarian endometriosis, deep infiltrating endometriosis.
Variations in urinary concentration phthalate metabolite levels in women with different symptoms of the disease | 24 months
  to evaluate potential variations in the levels of urinary phthalate metabolite in endometriosis patients in relation to the presence and levels of pain symptoms (dysmenorrhea, chronic pelvic pain, deep dyspareunia) and/or infertility.
Identify possible routes of exposure in everyday life and/or working environments | 24 months
  to evaluate potential confounders
Identify work context in which health risks for women could be highly than for men | 24 months
  to evaluate potential factors related to work context

CONTACTS AND LOCATIONS:
Overall Officials: Laura Buggio, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No